CLINICAL TRIAL: NCT01621867
Title: A Randomised, Double-blind, Placebo-controlled Phase 2B Clinical Trial of Repeated Application of Gene Therapy in Patients With Cystic Fibrosis
Brief Title: Repeated Application of Gene Therapy in CF Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Edinburgh (Other); University of Oxford (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ICL/CRO-1881; 2011-004761-33 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2012-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Gene therapy; CFTR gene; Gene expression; Non-viral; Multi dose
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pGM169/GL67A (CFTR Gene/Lipid Vector) (Active Comparator)
  Interventions: Drug: pGM169/GL67A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pGM169/GL67A — 5ml Gene Product/Lipid Vector pGM169/GL67A nebulised; 2ml nasal application of pGM169/GL67A in addition to 5ml nebulised gene product (Nasal Subgroup)
  Arms: pGM169/GL67A (CFTR Gene/Lipid Vector)
Drug: Placebo — 5ml Nebulised non-active placebo; 2ml nasal administration of non-active placebo (nasal subgroup)
  Arms: Placebo

SUMMARY:
Cystic fibrosis is a genetic condition where epithelial cells, including from the respiratory tract, have an abnormal function of a surface protein, the cystic fibrosis transmembrane conductance regulator (CFTR) protein resulting from abnormal gene expression. The trial will assess the clinical efficacy, safety & tolerability and gene expression following repeated nebulised doses of a gene product coding for a normal CFTR protein, with the primary outcome of the trial assessing lung function.

DETAILED DESCRIPTION:
Cystic fibrosis (CF), a common, genetically inherited disease, is caused by mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. This gene encodes the CFTR protein, which is expressed on the apical surface of epithelial cells, and which has many functions, the most important of which is thought to be ion transport. Abnormal ion transport leads to thick secretions in the airways, infection, inflammation and eventually irreversible lung damage. There is currently no treatment that halts the natural progression of the disease; all available successful therapies merely slow the rate of decline in clinical condition.

To date, no viral gene transfer agents retain efficacy upon repeated administration. Our study will assess the safety and efficacy of a lipid-mediated vector harbouring a normal CFTR gene in repeated nebulised administrations. We have completed a single dose safety study which evaluated the safety and gene expression of a single dose of pGM169/GL67A administered to the nose and lung of individuals with cystic fibrosis.

This trial is will randomise 130-patients to receive either a gene product (pGM169/GL67A)encoding for CFTR or placebo in a double-blinded fashion. All subjects will receive 12 doses of nebulised gene therapy at intervals of 4 weeks over a 48 week period. After dose 12 there will be 2 formal follow up visits, at 14 and 28 days post-dose. In addition, patients will be followed up long-term.

Subgroups of patients will be enrolled for gene expression measurement in both nose (at least n=20) and lower airway via bronchoscopy (at least n=20).

The primary outcome of the trial is to evaluate the relative change in predicted Forced Expiratory Volume in 1-second (FEV1) after 12-doses. Secondary outcome measures will assess the efficacy of the gene product (by assessment of patients' physiological function, serological indices, radiological appearances of the lungs and self-reported assessment of quality of life), on the degree of gene expression and on the product safely.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic fibrosis confirmed by sweat testing or genetic analysis
2. Males and females aged 12 years and above
3. Forced expiratory volume in the 1st second (FEV1) between 50 & 90% predicted inclusive (Stanojevic reference equations).
4. Clinical stability at screening defined by:

   1. Not on any additional antibiotics (excluding routine, long-term treatments) for the previous 2 weeks
   2. No increase in symptoms such as change in sputum production/colour, increased wheeze or breathlessness over the previous 2 weeks
   3. No change in regular respiratory treatments over the previous 4 weeks
   4. If any of these apply, entry into the study can be deferred
5. Prepared to take effective contraceptive precautions for the duration of their participation in the study and for 3 months thereafter (as stated in GTAC guidelines)
6. If taking regular rhDNase (pulmozyme) is willing, and considered able by independent medical carers, to withhold treatment for 24 hours before and 24 hours after the gene therapy dose (nebulised doses only)
7. Written informed consent obtained
8. Permission to inform their general practitioner of participation in study

Exclusion Criteria:

1. Infection with Burkholderia cepacia complex organisms, MRSA or M. abscessus
2. Significant nasal pathology including polyps, clinically-significant rhinosinusitis, or recurrent severe epistaxis (nose bleeds) (nasal cohort only)
3. Chloride secretory response on nasal PD of > 5 mV (nasal cohort only; will only be known after first measurement)
4. Acute upper respiratory tract infection within the last 2 weeks (entry can be deferred)
5. Previous spontaneous pneumothorax without pleurodesis (bronchoscopic subgroup only)
6. Recurrent severe haemoptysis (bronchoscopic subgroup only)
7. Current smoker
8. Significant comorbidity including:

   1. Moderate/severe CF liver disease (varices or significant, sustained elevation of transaminases: ALT/ AST>100 IU/l)
   2. Significant renal impairment (serum creatinine > 150 mmol/l)
   3. Significant coagulopathy (bronchoscopic group only)
9. Receiving 2nd line immunosuppressant drugs such as methotrexate, cyclosporine, intravenous immunoglobulin preparations
10. Pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Relative change in percent predicted FEV1 after 12 doses of gene product | 12-months

SECONDARY OUTCOMES:
EFFICACY | 12-months
  Relative change in other spirometric measures; lung clearance index; chest CT scan; Quality of Life Questionnaires; exercise capacity; activity monitoring; serum calprotectin; sputum culture; sputum weight, cell counts and inflammatory markers; frequency of antibiotics for increased chest symptoms
SAFETY | 12-months
  The above efficacy measures; clinical examination; transcutaneous oxygen saturation; serum inflammatory markers (CRP, white blood cell count,cytokines); renal and hepatic function; gas transfer; immune response markers (anti-nuclear and double-stranded DNA antibodies, CFTR-specific T cell responses); endobronchial histology (subgroup only)
GENE EXPRESSION(subgroups only) | 12-months
  Transgene mRNA expression in nasal and lower airway brushing samples; potential difference measurements in nose and bronchi.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Alton, MD, FMedSci, Study Director — Imperial College London; Jane Davies, MD, Principal Investigator — Imperial College London; Uta Griesenbach, PhD, Principal Investigator — Imperial College London; Steve Hyde, MA, DPhil, Principal Investigator — University of Oxford; Deborah Gill, PhD, Principal Investigator — University of Oxford; Chris Boyd, PhD, Principal Investigator — Edinburgh University; David Porteous, FMedSci, Principal Investigator — Edinburgh University; Alastair Innes, PhD, Principal Investigator — Edinburgh University; Steve Cunningham, PhD, Principal Investigator — Edinburgh University
Locations (3):
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Brompton Hospital, London

REFERENCES:
- [Result] Alton EW, Stern M, Farley R, Jaffe A, Chadwick SL, Phillips J, Davies J, Smith SN, Browning J, Davies MG, Hodson ME, Durham SR, Li D, Jeffery PK, Scallan M, Balfour R, Eastman SJ, Cheng SH, Smith AE, Meeker D, Geddes DM. Cationic lipid-mediated CFTR gene transfer to the lungs and nose of patients with cystic fibrosis: a double-blind placebo-controlled trial. Lancet. 1999 Mar 20;353(9157):947-54. doi: 10.1016/s0140-6736(98)06532-5. PMID 10459902
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818
- [Derived] Alton EWFW, Armstrong DK, Ashby D, Bayfield KJ, Bilton D, Bloomfield EV, Boyd AC, Brand J, Buchan R, Calcedo R, Carvelli P, Chan M, Cheng SH, Collie DDS, Cunningham S, Davidson HE, Davies G, Davies JC, Davies LA, Dewar MH, Doherty A, Donovan J, Dwyer NS, Elgmati HI, Featherstone RF, Gavino J, Gea-Sorli S, Geddes DM, Gibson JSR, Gill DR, Greening AP, Griesenbach U, Hansell DM, Harman K, Higgins TE, Hodges SL, Hyde SC, Hyndman L, Innes JA, Jacob J, Jones N, Keogh BF, Limberis MP, Lloyd-Evans P, Maclean AW, Manvell MC, McCormick D, McGovern M, McLachlan G, Meng C, Montero MA, Milligan H, Moyce LJ, Murray GD, Nicholson AG, Osadolor T, Parra-Leiton J, Porteous DJ, Pringle IA, Punch EK, Pytel KM, Quittner AL, Rivellini G, Saunders CJ, Scheule RK, Sheard S, Simmonds NJ, Smith K, Smith SN, Soussi N, Soussi S, Spearing EJ, Stevenson BJ, Sumner-Jones SG, Turkkila M, Ureta RP, Waller MD, Wasowicz MY, Wilson JM, Wolstenholme-Hogg P; UK Cystic Fibrosis Gene Therapy Consortium. Repeated nebulisation of non-viral CFTR gene therapy in patients with cystic fibrosis: a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Respir Med. 2015 Sep;3(9):684-691. doi: 10.1016/S2213-2600(15)00245-3. Epub 2015 Jul 3. PMID 26149841
- See also: The UK Cystic Fibrosis Gene Therapy Consortium — http://www.cfgenetherapy.org.uk/